CLINICAL TRIAL: NCT01624324
Title: Aminoglycoside Plasma Level Measurement in Neonates With Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Rianto Setiabudy, Prof. Dr. dr. SpFK(K), Indonesia University
Other Study IDs: Aminoglycoside
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Nephrotoxicity; Ototoxicity
Keywords: aminoglycoside; KIM-1; DPOAE; nephrotoxicity; ototoxicity
MeSH Terms: conditions — Ototoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Plasma, Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine whether the plasma concentration of aminoglycoside in Indonesia neonates with infection are within safe and effective range and its association with cochlear toxicity and nephrotoxicity.

DETAILED DESCRIPTION:
Aminoglycosides are toxic antibiotics, but they are urgently needed to treat newborns with severe infections. Aminoglycosides are well known for their nephrotoxicity and ototoxicity, meanwhile the renal function of the newborns is not yet fully developed.The aminoglycoside dosage currently applied in Indonesia is derived from studies done in Caucasian populations. The safety and efficacy of this dosage regimen, however, have never been evaluated till date. The pharmacokinetic profile of drugs may vary between populations and this may be influenced by genetic factors, lifestyle, drug interactions, etc. The detection of aminoglycoside toxicity in newborns is usually problematic. The present study aims to know the proportion of nephrotoxicity and ototoxicity in newborns in the Cipto Mangunkusumo Hospital treated with gentamicin or amikacin in relation to their trough serum concentration. The serum level of gentamicin and amikacin is assumed to be safe if the trough serum concentrations are < 2 mcg/mL and effective if its is between 5-12 mcg/mL. For amikacin the desired trough serum concentrations are <10 mcg/mL and the peak is between 20-30 mcg/mL. The nephrotoxicity was assessed by measuring the level of kidney injury molecule-1 in urine while the ototoxicity was assessed by Distortion Product Otoacoustic Emission (DPOE) instrument.

ELIGIBILITY:
Inclusion Criteria:

* neonates with infection treated with gentamicin or amikacin

Exclusion Criteria:

* neonates who hypersensitive to gentamicin and amikacin
* neonates who also treated with other nephrotoxic drugs (vancomycin, furosemide, amphotericin B, meropenem)

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates hospitalized in Perinatology Division, Pediatric Department, Cipto Mangunkusumo Hospital with severe infection requiring an aminoglycoside therapy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2010-11

CONTACTS AND LOCATIONS:
Locations (1):
- Perinatology Division, Pediatric Department, Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Derived] Setiabudy R, Suwento R, Rundjan L, Yasin FH, Louisa M, Dwijayanti A, Simanjuntak E. Lack of a relationship between the serum concentration of aminoglycosides and ototoxicity in neonates. Int J Clin Pharmacol Ther. 2013 May;51(5):401-6. doi: 10.5414/CP201833. PMID 23557866